CLINICAL TRIAL: NCT04055142
Title: A Phase III, Randomized, One-site, Pilot, Open-label, Parallel Groups Trial for Evaluating the Efficacy and Safety of Electrocoagulation vs Topic Sinecatechins vs Topic Cidofovir Within the Treatment to High-grade Anal Intraepithelial Neoplasia in HIV Homosexual Males
Brief Title: Clinical Trial for Evaluating the Efficacy and Safety of Electrocoagulation vs Topic Sinecatechins vs Topic Cidofovir Within the Treatment to High-grade Anal Intraepithelial Neoplasia in HIV Homosexual Males
Acronym: TreatAIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TreatAIN
Record Dates: First submitted 2019-07-19; First posted 2019-08-13 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: High-grade Anal Intraepithelial Neoplasia
MeSH Terms: interventions — Electrocoagulation; Cidofovir; Ointments; green tea extract polyphenone E

STUDY DESIGN:
Intervention Model Description: A phase III, randomized, one-site, pilot, open-label, parallel groups trial for evaluating the efficacy and safety of electrocoagulation vs topic sinecatechins vs topic cidofovir within the treatment to high-grade anal intraepithelial neoplasia in HIV homosexual males.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Electrocoagulation (Active Comparator): This procedure will be implemented following the Standard of Care (SoC) on weeks: 0, 8 and 16 calculated since the day the patient is included into the trial.
  Interventions: Procedure: electrocoagulation
- Sinecatechins (10%) (Experimental): Topical ointment wich contains 2 grams of active principle (sinecatechins 10%) at each administration. It will be taken three times per week during 8 weeks of treatment.
  Interventions: Drug: sinecatechins 10% topical ointment
- cidofovir (1%) (Experimental): Topical ointment wich contains 2 grams of active principle (cidofovir 1%) at each administration. It will be taken three times per week during 8 weeks of treatment.
  Interventions: Drug: cidofovir 1% topical ointment

INTERVENTIONS:
Procedure: electrocoagulation — HIV homosexuals males with High-grade anal intraepithelial neoplasia will be randomized and electrocoagulation will be performed in 2-3 sessions (session every 2 weeks)
  Arms: Electrocoagulation
Drug: cidofovir 1% topical ointment — HIV homosexuals males with High-grade anal intraepithelial neoplasia will be randomized and they will be treated with cidofovir 1% ointment (3 times per week during 8 weeks)
  Other Names: Cidofovir
  Arms: cidofovir (1%)
Drug: sinecatechins 10% topical ointment — HIV homosexuals males with High-grade anal intraepithelial neoplasia will be randomized and they will be treated with sinecatechins 10% ointment (3 times per week during 8 weeks)
  Other Names: Veregen ointment
  Arms: Sinecatechins (10%)

SUMMARY:
This study wants to demonstrate the non-inferiority in terms of efficacy and safety of treatment with cidofovir (1%) in topical ointment or topical sinecatechins (10%) ointment versus electrocoagulation (control group) for the treatment of high-grade anal intraepithelial neoplasia (HGAIN).

The target patients are Human Immunodeficiency Virus (HIV)-infected homosexual males.

All these patients will be randomized by a proportion of 1:1:1 setting up 3 different parallel arms of the study: control group, cidofovir (1%) group and topical sinecatechins (10%) group.

DETAILED DESCRIPTION:
This Trial addresses one of the emerging problems in patients with HIV infection, such as the high incidence of anal dysplasia and anal cancer. The study proposes to evaluate new therapeutic options in the treatment of anal dysplasia, thus trying to overcome the current limitations of electrocoagulation (moderate efficacy, high recurrence, significant patient discomfort, and significant health cost).

Topical cidofovir has shown (in a non-comparative study) efficacy and tolerance rates similar to those observed for electrocoagulation, although with the benefits of self-application by the patient. This makes it an attractive topical treatment option that requires a direct comparison with the currently chosen treatment, which is electrocoagulation.

On the other hand, the medical properties of the sinecatechins, together with the results obtained in the treatment studies of oral and cervical dysplasia, and the possibility of being self, make this drug an attractive option to be evaluated experimentally in the treatment of anal dysplasia. Finally, the identification of prognostic markers of the disease should continue to be explored, in terms of the response to treatment and the recurrence of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Men who have sex with men, older or same than 18 years old.
* HIV-1 positive men.
* High grade anal intraepithelial neoplasia recognised by biopsy during 12 months previous to study.
* Informed consent is signed voluntarily.

Exclusion Criteria:

* Patient with any disease or condition which rules him out to participate in the research, by investigator opinion.
* Treated patients for HGAIN in the previous 6 months.
* Patients with relapsed HGAIN two or more times in the last three months.
* People with learning difficulties

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-07-02 (Actual)

PRIMARY OUTCOMES:
% of patients with complete or partial regression of high grade anal intraepithelial neoplasia (HGAIN) at 10 weeks after end of treatment (with a permitted deviation of 4 weeks). | 10 weeks
  % of patients with complete or partial regression of high grade anal intraepithelial neoplasia (HGAIN) at 10 weeks after end of treatment (with a permitted deviation of 4 weeks).
  sinecatechins 10% ointment treatment for high grade anal intraepithelial neoplasia (HGAIN) with respect to electrocoagulation treatment in HIV-positive men who have sex with men.

SECONDARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as assessed by CTCAE v4.0 during the study. | 48 weeks
  By monitoring activities related with pharmacovigilance duties during the patient participation of each patient.
Number of Participants With analytical and clinical Adverse Events as assessed by CTCAE v4.0 during the study. | 48 weeks
  To describe the proportion of clinic and laboratory adverse events, which imply treatment dropout, in research treatment arm especially (cidofovir and sinecatechins). By monitoring activities related with pharmacovigilance duties during the patient participation of each patient
Median score obtained in the HIV Treatment Satisfaction Questionnaire (HIVTSQ). | 48 weeks
  HIVTSQ has been modified by replacing the references to "HIV treatment" with "anal dysplasia treatment", and eliminating question 2 of HIVTSQ.
  The following questions are related to the treatment you are being given in the trial and your experience in recent weeks. Please answer each question by circling a number on each of the scales evaluating them from 6 (very satisfied) to 0 (not satisfied).
  * To what extent are you satisfied with your current treatment?
  * To what extent are you satisfied with the side effects you have had from your current treatment?
  * To what extent are you satisfied with the requirements related to your current treatment?
  * To what extent do you consider your treatment to be comfortable / practical?
  * o what extent do you think your treatment is flexible?
  * To what extent are you satisfied with the information / knowledge you have about anal dysplasia?
  * To what extent are you satisfied with the degree to which the treatment adapts to your
% of patients who reduce the measurement in HGAIN octants, although without regression, by high-resolution anoscopy at 10 weeks after end of treatment (with a permitted deviation of 4 weeks). | 10 weeks (+/- 4 weeks) after end of treatment
  To compare % of decreased extension of HGAIN patients, with absence of regression during the study period according to protocol schedule.
% of patients with no Human Papilloma Virus(HPV) detection at 10 weeks after end of treatment (with a permitted deviation of 4 weeks). | 10 weeks (+/- 4 weeks) after end of treatment
  To compare % of Human Papilloma Virus clearance in patients during the study period according to protocol schedule.
Number of participants with a new HGAIN at histological sample after a complete or partial result after treatment | 48 weeks
  During the study period according to protocol schedule.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital U. Vall d'Hebrón, Barcelona, Catalonia, Spain

REFERENCES:
- [Derived] Burgos J, Curran A, Garcia J, Campany D, Descalzo V, Suanzes P, Navarro J, Planas B, Sanchiz M, Landolfi S, Dinares C, Hernandez-Losa J, Falco V. Effectiveness of Electrocautery, Topical Cidofovir, and Topical Sinecatechins for the Treatment of Anal High-Grade Squamous Intraepithelial Lesions in Persons With HIV: An Open-Label, Randomized Controlled Trial. Clin Infect Dis. 2025 Sep 16;81(2):333-340. doi: 10.1093/cid/ciaf086. PMID 40036375